CLINICAL TRIAL: NCT05909020
Title: EVolution of a patiEnt-REported Symptom-based Risk Stratification sySTem to Redesign the Suspected Head and Neck Cancer Referral Pathway (Phase 1)
Brief Title: EVEREST-HN 1: EVolution of a patiEnt-REported Symptom-based Risk Stratification sySTem
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5683
Record Dates: First submitted 2023-05-09; First posted 2023-06-18 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Approximately 150 adults referred for suspected HNC will be recruited.
  Interventions: Other: No intervention.
- Staff: Approximately 15 ENT and Maxillofacial) clinicians will be recruited.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — No intervention.

SUMMARY:
Can a patient-reported symptom-based risk stratification system improve the suspected head and neck cancer (HNC) pathway?

Our methodology includes six interlinked work packages to deliver our aim, with EVEREST-HN 1 encompassing the first of these and seeking to optimise a patient-reported symptom inventory for HNC and outline requirement specification for the SYmptom iNput Clinical (SYNC) system.

DETAILED DESCRIPTION:
The EVEREST-HN pathway should be based on a comprehensive understanding of existing HNC diagnostic pathways and what patients and clinicians value in these. The language used within the EVEREST pathway needs to be accessible and optimal to elicit appropriate information.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Adults ≥ 18 years referred via suspected HNC pathway without previous history of HNC
* Participants willing and able to give informed consent for participation in the study.

Clinicians:

* Staff at participating sites involved in the diagnostic pathway for people with suspected HNC.

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Recruitment will aim for variation in age, ethnicity, socio-economic status, presenting symptoms.
  Clinicians Clinical staff involved in HNC diagnosis. Varying in seniority (consultant, registrar) and specialty (ENT, maxillofacial)
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Inventory and specification for the SYmptom iNput Clinical (SYNC) system | September 2022 - August 2023
  To optimise a patient-reported symptom inventory for HNC and outline requirement specification for the SYmptom iNput Clinical (SYNC) system

SECONDARY OUTCOMES:
To further explore the current suspected HNC pathway and the language used when discussing symptoms. | September 2022 - August 2023
  To understand how clinicians decide subsequent steps for patients referred with suspected HNC, the language patients and clinicians use to describe symptoms and patients' and clinicians' views and experiences of the current diagnostic process for HNC. with a focus on what would work for EVEREST-HN study.

CONTACTS AND LOCATIONS:
Overall Officials: Vinidh Paleri, Study Chair — Royal Marsden NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Luton & Dunstable University Hospital, Luton
  - Oxford NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No